CLINICAL TRIAL: NCT05696002
Title: Advanced Pelvic Surgical Oncology Database - Prospective Observational Study
Status: Recruiting | Type: Observational
Sponsor: Glasgow Royal Infirmary (Other)
Responsible Party: Principal Investigator, Norman Galbraith, NES/CSO Clinical Lecturer in Surgery, Glasgow Royal Infirmary
Other Study IDs: APSOD
Record Dates: First submitted 2023-01-10; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Rectal Cancer; Pelvic Cancer; Gynecologic Cancer; Colon Cancer
Keywords: Pelvic exenteration; Abdominoperineal resection; Reconstructive flap; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms; Pelvic Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Not currently, but in the future, plans to study circulating immune cell/cytokine measurements, ctDNA, peritoneal macrophage/neutrophils, and existing protocols for biobanking of tumour samples/organoids
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced pelvic oncological resection: Complex resection

SUMMARY:
Retrospective and prospective observational study of patients undergoing advanced pelvic oncological resection for maligancy including multi visceral resection, beyond TME resection and sacrectomy/flap reconstruction/urinary reconstruction at Glasgow Royal Infirmary.

Goal is to study and report outcomes for patients to characterise and understand major complications, natural history of resectional patients and identify areas for future interventional study.

DETAILED DESCRIPTION:
Retrospective and prospective observational study of patients undergoing advanced pelvic oncological resection for maligancy including multi visceral resection, beyond TME resection and sacrectomy/flap reconstruction/urinary reconstruction at Glasgow Royal Infirmary.

Goal is to study and report outcomes for patients to characterise and understand major complications, natural history of resectional patients and identify areas for future interventional study..

ELIGIBILITY:
Inclusion Criteria:

* Advanced pelvic oncological resection defined as more than 1 pelvic organ resected

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tertiary referral centre
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-14 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Cancer-specific survival | 10 years
  Months
Overall survival | 10 years
  Months
Post-operative complications | 10 years
  Frequency
Quality of life (survey) | 10 years
  Score

CONTACTS AND LOCATIONS:
Overall Officials: Colin Steele, PhD FRCS, Study Director — Glasgow Royal Infirmary
Locations (1):
- Academic Department of Surgery, Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided